CLINICAL TRIAL: NCT04066465
Title: Neurocognitive Function /executive Functions After Proton Therapy in Children and Adolescents.
Brief Title: Neurocognitive Function After Proton Therapy in Children and Adolescents
Acronym: ELBE-ProKids
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Gert und Susanna Mayer Stiftung (Unknown)
Responsible Party: Sponsor
Other Study IDs: STR-ELBE-Pro-Kids-2019
Record Dates: First submitted 2019-06-19; First posted 2019-08-26 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Primary Brain Tumor
Keywords: Brain Tumor; children and adolescents; neurocognitive function; neurocognitive or neuropsychological outcome; quality of life, LOQ; EEG; Neuropsychological Tests; Proton Therapy; Neurosurgical Treatment
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Proton Therapy: Patients receive proton Radio(chemo)therapy according to clinical standard. Proton Treatment is indicated BEFORE inclusion into the trial ans is not part of the trial. Neurological status and neurocognitive testing on core executive functions (inhibition, working memory, cognitive flexibility) and Quality of life measurements are performed regularely during follow-up using standardized KINDL® questionnaires for general quality of life and specific for oncologic diseases. In addition to the treatment parameters of the radio(chemo)therapy protocol, further radiation doses to brain substructures and organs at risk are documented.
- No Radiotherapy - Surgical only group: Patients are included AFTER surgery of their brain tumour and receive no radiotherapy due to their disease (i.e. according to clinical standard). This Treatment is not part of the trial, but stratifies the Patient in this second Group.
  Neurological status and neurocognitive testing on core executive functions (inhibition, working memory, cognitive flexibility) and Quality of life measurements are performed regularely during follow-up using standardized KINDL® questionnaires for general quality of life and specific for oncologic diseases.
- Control Group: Healthy kids are recruited as Standard Group.
  Neurological status and neurocognitive testing on core executive functions (inhibition, working memory, cognitive flexibility) and Quality of life measurements are performed regularely using standardized KINDL® questionnaires for general quality of life and specific for oncologic diseases.

SUMMARY:
Brain tumors are the second most frequent malignant diseases in children and adolescents. In the study the short and medium term consequences of proton therapy on cognitive processes in particular on executive functions in pediatric patients shall be highlighted/analysed/evalutated. In a second step, these results are to be compared with

1. a group of children and adolescents who had only /exclusively had operative therapy and
2. with a healthy control group. Thus, the extent to which these treatment options differ in terms of their short and medium-term effect is assessed. Methods of neurocognitive/neurophysiology brain research approaches are applied that may potentially visualize even small / subtle changes in mental activities/neurocognitive function. Therefore the effects of treatment can be evaluated and the neuropsychological outcome of children and adolescents with brain tumors can be improved.

DETAILED DESCRIPTION:
Radio(chemo)therapy with protons is conducted according to current treatment standards or, for patients participating in a clinical intervention study, according to the study protocols of the GPOH. Only patients with prescribed radiation doses > 40 Gy (RBE) will be included. Treatment planning, the target volume and radiotherapy will be performed according to the current treatment standards. For patients participating in a clinical intervention study, radiotherapy is corresponding to study protocol of the GPOH. Risk organs (e.g. brain stem, chiasma, optic nerves, gll. Lacrimals, lenses, inner ears and spine) are contoured and the radiation doses for these organs are limited according to institutional guidelines. Radiotherapy is performed according to guidelines, i.e. 5 days a week for 4-6 weeks, usually on an outpatient basis.

ELIGIBILITY:
Indication: Patients with primary brain tumor

Inclusion Criteria:

* all groups: Patients in childhood and adolescence between 8-18 years of age
* all groups: no prior radiotherapy of the brain,
* all groups: The patient is able to perform repeated neuropsychological tests (approx. 1 hour per examination),
* all groups: corrected visual acuity not impaired below 80% or no subjective indication of visual acuity impairment,
* all groups: corrected hearing not impaired or no subjective evidence of hearing impairment,
* all groups: Patient is able to perform follow-up examinations,
* all groups: written consent of the patient/parent or guardian.
* Brain tumour groups with/without irradiation: Primary brain tumour
* brain tumor groups with/without radiation: curative or long-term palliative intention of therapy
* brain tumor groups with/without irradiation: life expectancy > 3 years
* Irradiation group only: planned proton therapy with a local radiation dose of at least 40 Gy(RBE)

Exclusion Criteria:

* Patients under 8 or over 18 years of age (We limit the study to children over 8 years of age due to the fact that executive functions mature very late.)
* Brain metastases from extracerebral tumors
* Patient receives intrathecal chemotherapy
* pure palliative treatment concept
* The patient is not able to perform repeated neuropsychological tests (approx. 1 hour per examination).
* Chronic diseases that may affect the results of neurological EEG and neuropsychological examinations.
* The patient is not in a position to perform follow-up examinations
* no written consent of the patient / parent or legal guardian
* Participation in an intervention study whose procedures contradict those of the present study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 30 patients with infra-tentorial or supra-tentorial tumors undergoing proton therapy, 30 patients undergoing surgical treatment and a control cohort of 30 adolescents. Therefore, a total of 90 persons will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological correlates of cognitive control (ERP amplitude measures, spectral power measures) | 2 years
  Neurophysiological processes are examined while subjects perform the cognitive tests.
Quality of Life Parameters (KINDL®) | 2 years
  QoL Parameters are measured and reported using KINDL® questionnaires for general quality of life and specific for oncologic diseases (also KINDL®). Scales for QoL items are 0-100 (with 100 being the Optimum, i.e. lower values indicating worse outcome). Evaluation is performed according to the standard published with the validated questionnaires (https://www.kindl.org/deutsch/fragebögen/)

SECONDARY OUTCOMES:
dose-volume parameters to normal tissues, i.e. maximum irradiation doses, mean doses and doses to subvolumes | 2 years
  physical doses to substructures of the brain are collected and correlated with neurophysiological outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Mechthild Krause, Prof. Dr., Study Chair — University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology, German Consortium for Translational Cancer Research (DKTK)
Locations (3):
- Germany (3):
  - University Hospital Carl GUstav Carus Dresden, Child and adolescent psychiatry and psychotherapy, Dresden, Saxony
  - University Hospital Carl GUstav Carus Dresden, Department of Neuropaediatrics, Dresden, Saxony
  - University Hospital Carl GUstav Carus Dresden, Department of Radiation Therapy and Radiation Oncology, Dresden, Saxony

IPD SHARING:
Plan to Share IPD: No